CLINICAL TRIAL: NCT00626054
Title: Comparison of Two Methods of Administration of a PEG Solution During Bowel Preparation for Colonoscopy in Hospitalized Patients
Brief Title: Comparison of Two Methods of Administration of a PEG Solution
Acronym: PEG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Ram Dickman, Gastroenterology Institute Deputy-manager, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004907
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Colorectal Cancer
Keywords: Colonoscopy; PEG Solution
MeSH Terms: conditions — Colorectal Neoplasms | interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Group 1 will receive the precolonoscopy PEG solution in a single dose of 3 liters in the evening preceding the test.
  Interventions: Drug: PEG solution in a single dose of 3 liters
- 2 (Active Comparator): Group 2 will receive half the dose (1.5 liters) of the identical solution in the evening preceding the test and the other half (1.5 liters) on the morning of the test.
  Interventions: Drug: PEG solution

INTERVENTIONS:
Drug: PEG solution in a single dose of 3 liters — Group 1 will receive the precolonoscopy PEG solution in a single dose of 3 liters in the evening preceding the test.
  Other Names: Meroken New
  Arms: 1
Drug: PEG solution — PEG solution: half the dose (1.5 liters) of the identical solution in the evening preceding the test and the other half (1.5 liters) on the morning of the test
  Other Names: Meroken New
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness (quality of bowel cleansing) and ease of use (patient satisfaction) of two methods of administration of a precolonoscopy PEG solution in hospitalized patients.

DETAILED DESCRIPTION:
Background and rationale of the research

Colonoscopy is an endoscopic examination whereby the physician can visually inspect the interior lining of the colon. It is the most efficient and accurate means of identifying, either directly or by biopsy, neoplasms in the large intestine and inflammatory processes, infections, or ischemia involving the whole colon and the distal small intestines. In addition, during the procedure, certain endoscopic treatments may be performed, such as removal of precancerous polyps and cauterization of bleeding sites such as vascular malformations by electrocoagulation.

Proper preparation of the bowel prior to colonoscopy is crucial to the quality of the examination. Suboptimal preparation can adversely affect the ability of the examiner to detect abnormalities in the small and large intestine or to carry out various endoscopic treatments. In some cases, poor preparation may necessitate canceling the procedure and rescheduling the patient for a repeated test.

To properly clear the bowel, patients must strictly adhere to a special diet and drink a laxative solution as directed. The physician selects the specific type of laxative solution from among those that are currently available on the basis of the patient's age and underlying diseases. At present, polyethylene glycol (PEG), owing to its good safety profile and relative lack of complications, is recommended in older patients (65 years or more), patients with hypertension or renal or cardiac insufficiency, and patients being treated with diuretics and ACE inhibitors. However, a major disadvantage of PEG is its difficulty of use, which involves bad taste and drinking 3 liters within a short period of time on the day before the examination.

Several recent studies in the medical literature have reported that in ambulatory patients, dividing the oral laxative solution into 2 doses taken at different times is more effective than drinking the whole amount in one session. On the basis of these findings, and given that the quality of the bowel preparation is known to be poorer in hospitalized than in ambulatory patients, we sought to determine if dividing the laxative dose will yield better results in hospitalized patients as well. It should be noted that laxative solutions constitute the most accepted method of preparing the bowel for colonoscopy and that in the present study, the sole difference from standard practice was the method of administration, namely a single or a split dose.

Aim of the study The purpose of this study is to compare the effectiveness (quality of bowel cleansing) and ease of use (patient satisfaction) of two methods of administration of a precolonoscopy PEG solution in hospitalized patients.

Method

Study design: Prospective, comparative, randomized

End points:

Primary - Cleanliness of the bowel, as determined by the examiner, and ease of use, as determined by a patient satisfaction questionnaire in the two study arms Secondary - Effect of external factors (demographic parameters, length of hospitalization, procedural diagnosis) on the quality of the bowel preparation.

Study sample: Four hundred hospitalized patients scheduled for a colonoscopy examination as part of their in-hospital work-up.

Inclusion criteria: Age 18-80 years; ability to understand and complete the questionnaires; ability to participate in all stages of the research.

Exclusion criteria: Previous colon surgery, previous endoscopic procedures under full anesthesia, known sensitivity to the PEG solution, terminal renal or cardiac insufficiency, inability to sign the informed consent form Colonoscopy: All patients will perform the precolonoscopy bowel preparation by one of two methods, according to the study design, followed by colonoscopy at the Gastrolenterology Institute of Rabin Medical Center

Questionnaires:

Demographic questionnaire - age, sex, weight, height, years of education Patient satisfaction questionnaire - ease of preparation and related symptoms In addition, physicians will rate the degree of bowel visibility after the procedure on a standard scale.

Study design:

The study sample will include hospitalized patients scheduled for colonoscopy. The physicians conducting the research will obtain informed consent from all candidates for the study prior to their enrollment.

At onset of the study, the participants will complete a demographic questionnaire in the presence of a member of the research team. Items will include age, sex, height, weight, and years of education.

Study participants will be randomly divided into 2 groups. Group 1 will receive the precolonoscopy PEG solution in a single dose of 3 liters in the evening preceding the test. Group 2 will receive half the dose (1.5 liters) of the identical solution in the evening preceding the test and the other half (1.5 liters) on the morning of the test. The randomization will be performed at the Gastroenterology Institute. The secretary of the Institute will then inform the nurses/attendants in the various hospitalization departments which of the two procedures to apply to each individual patient. Before the procedure, the patients will complete a demographic questionnaire in the presence of a member of research team. The physician performing the colonoscopies will be blinded to the group allocation. After completing the colonoscopy, the physician will rate the quality of the bowel preparation in the patient's medical file according to the Aronchick scale, as follows:

Score Description 0 - excellent More than 95% of the intestines visible

1. - good Large amount of transparent fluid requiring suction; more than 90% of intestines visible
2. - fair Semisolid stool requiring suction/flushing; more than 90% of intestines visible
3. - poor Semisolid stool difficult or impossible to remove; less than 90% of intestines visible
4. - failed Repeated test required

Following the procedure, study participants will be asked to rate their satisfaction with the ease of use of the bowel preparation and the severity of symptoms related to it (e.g., stomach pain, nausea) on a VAS scale.

Colonoscopy method:

At the time of referral for colonoscopy, patients will receive a preliminary explanation of the test, of the alternative examinations currently available, and of any possible complications of the test. On the day of the colonoscopy, after receiving additional explanations from the attending gastroenterologist, patients will be asked to sign an informed consent form. The colonoscopy examination will be performed with patients lying on their left side; a sedative will be administered intravenously. During the procedure, the patient may feel cramping and discomfort from the infusion of air into the colon. The duration of the examination will about 30 minutes, depending on the structure of the colon, the amount of visibility consequent to the bowel preparation, and the degree of patient cooperation; the last two factors are essential for the success of the procedure. The endoscopic device will be carefully cleaned and sterilized between examinations in accordance with routine practice at our institute and accepted standards in developed countries.

Statistical analysis

On the basis of reported means and standard deviations in the medical literature, assuming a 75% compliance rate and type 1 error (α) of 0.05, a study sample of 400 hospitalized patients will yield a statistical power of more than 80%. The sample will be divided into two treatment groups using the computerized Research Randomizer 2007 (http://www.randomizer.org/) Independent t test will be used to compare means of continuous variables between the two groups, and chi-square test will be used to compare proportions. Nonparametric Mann-Whitney test will be used to analyze the level of preparation and bowel cleanliness, ranked on an ordinal scale, between the groups. All test will be two-sided; statistical significance will be set at p<0.05. All analyses will be performed with SPSS software, version 15.

Participating researchers

Gastroenterology Institute: Dr. Ram Dickman, Dr. Gal Eyal, Dr. Zvidi Ibrahim, Dr. Ofer Ben Bassat, Dr. Wilkin Alexander, Dr. Zohar Levy, Dr. Michal Cohen, Dr. Gerald Fraser, Prof. Yaron Niv, Dr. Boris Sapoznikov, Dr. Irit Avni-Biran, Nechama Horev, Melli Mor, Negba Segal, Shlomit Flaut, Yafit Honen, Igor Bogoslavsky, Ilana Morad.

Schedule

The study is planned for a two-year period:

Patient enrollment until mid-2009 Data collection and analysis until end 2008-beginning 2009

Ethics

Patient anonymity will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* ability to understand and complete the questionnaires
* ability to participate in all stages of the research

Exclusion Criteria:

* Previous colon surgery
* endoscopic procedures under full anesthesia
* known sensitivity to the PEG solution
* terminal renal or cardiac insufficiency
* inability to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Cleanliness of the bowel, as determined by the examiner, and ease of use, as determined by a patient satisfaction questionnaire in the two study arms | 1 year

SECONDARY OUTCOMES:
Effect of external factors (demographic parameters, length of hospitalization, procedural diagnosis) on the quality of the bowel preparation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Niv, Prof, Study Director — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel